CLINICAL TRIAL: NCT05818800
Title: Pilot Study of Information and Communication Technology Solutions for Hypertension Care
Brief Title: Pilot Study Based on Technology Solutions for Hypertension Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 09E801
Record Dates: First submitted 2023-03-20; First posted 2023-04-19 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Hypertension; Blood Pressure
Keywords: Digital Technology; hypertension; blood pressure
MeSH Terms: conditions — Hypertension | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This will be a randomised controlled trial where patients with hypertension will be randomised either to one of the two digital solutions or to standard care.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Solution 1 - HSmartBPM (developed by a supplier consortium led by GNOMON) (Other): Solutions consist of devices (e.g., blood pressure monitors, body composition scales) working together in an ecosystem enabled by a user-facing service and associated interfaces. Users are invited to a dedicated training session at the pilot site to officially become enrolled and begin using the solution for an extended period of time. During that time, users are instructed to use the solutions based on recommendations by their treating physicians (e.g., regular measurement of blood pressure using the solution, or scheduling of regular visits via the solution interface). Questionnaires are administered via the solution's interface at the beginning and end of the trial duration. At the end of the trial, the user is asked to return the devices to the pilot site.
  Interventions: Device: digital solution
- Solution 2 - HyperHealth (developed by a supplier consortium led by TECH4CARE) (Other): Solutions consist of devices (e.g., blood pressure monitors, body composition scales) working together in an ecosystem enabled by a user-facing service and associated interfaces. Users are invited to a dedicated training session at the pilot site to officially become enrolled and begin using the solution for an extended period of time. During that time, users are instructed to use the solutions based on recommendations by their treating physicians (e.g., regular measurement of blood pressure using the solution, or scheduling of regular visits via the solution interface). Questionnaires are administered via the solution's interface at the beginning and end of the trial duration. At the end of the trial, the user is asked to return the devices to the pilot site.
  Interventions: Device: digital solution
- control (Other): the control group where they will be followed according to standard care
  Interventions: Other: Standard Care

INTERVENTIONS:
Device: digital solution — randomised controlled trial where patients with hypertension will be randomised either to one of the two digital solutions
  Arms: Solution 1 - HSmartBPM (developed by a supplier consortium led by GNOMON); Solution 2 - HyperHealth (developed by a supplier consortium led by TECH4CARE)
Other: Standard Care — randomised controlled trial where patients with hypertension will be randomised r to standard care
  Arms: control

SUMMARY:
The goal of this clinical trial is to understand whether the adoption of digital solutions by healthcare professionals and patients improves the management of patients with high blood pressure.

The main questions it aims to answer are:

* are these digital solutions feasible and well accepted by patients?
* can these solutions, compared to standard care, allow a better hypertension control in patients with high blood pressure?

Participants randomised to one of the two intervention arms will be asked to adopt the digital solutions that include a smartphone app and 2 devices for blood pressure and body weight measurement that will be connected to the app.

Researchers will compare patients randomised in the two intervention groups with patients randomised to standard care (control group)

DETAILED DESCRIPTION:
The study falls within the scope of the HSMonitor project, a pre-commercial tender for the development of telematics solutions aimed at optimising patient health status and disease management. Specifically, the aim of this study is to test whether the adoption of HSMonitor solutions by healthcare professionals and patients improves the management of patients with high blood pressure.

This will be a randomised controlled trial where patients with hypertension will be randomised either to one of the two digital solutions or to standard care.

The present pilot study is planned to be carried out within the framework of the EU project HSMonitor - Pre-commercial Procurement of innovative ICT-enabled monitoring to improve health status and optimize hypertension care (Grant Agreement Nr. 856698).

The two solutions are referred to as:

* Solution 1 - HSmartBPM (developed by a supplier consortium led by GNOMON)
* Solution 2 - HyperHealth (developed by a supplier consortium led by TECH4CARE)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with essential hypertension (>140/90 mmHg or normal BP with antihypertensive treatment)
* Basic ICT knowledge and ability to access the internet at home and on mobile devices
* aged 18+
* ability to provide written informed consent, giving informed consent.
* written informed consent

Exclusion Criteria:

* inability to consent
* chronic renal replacement therapy (haemodialysis, peritoneal dialysis or transplantation) or if, at baseline, there is a history of active malignancy within the last five years
* pregnancy
* illiterate
* younger than 18 years
* being a prisoner
* being institutionalized
* the patient is mentally or psychiatrically ill
* the patient has barriers to understand the implications of participation to the study
* the patient is critically ill or dying
* the patient is extremely poor
* the patient has a learning disability
* the patient is sedated or unconscious
* the patient is a refugee with no permanent permission to stay
* the patient does not have a good command of the language
* the patient has problems in cognitive, juridical, and deferential dimensions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-12-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in blood pressure | 2 and 6 months
  The changes in systolic and diastolic blood pressure

SECONDARY OUTCOMES:
The user satisfaction measured with VAS | 2 and 6 months
  0-100 points VAS where 0 means not satisfied and 100 fully satisfied

OTHER OUTCOMES:
Quality of life measured with EQ-5D | 2 and 6 months
  EQ-5D is a standardised measure of health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Parati, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Italy